CLINICAL TRIAL: NCT01548911
Title: Safety and Efficacy of Gemtuzumab Ozogamicin (Mylotarg®) as for Treatment of Patients With CD33-Positive Acute Myeloid Leukemia (AML)
Brief Title: Gemtuzumab Ozogamicin in Treating Patients With Acute Myeloid Leukemia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00019491; NCI-2012-00127 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 22311 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2012-02-14; First posted 2012-03-08 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Promyelocytic Leukemia (M3); Recurrent Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Congenital Abnormalities; Leukemia, Promyelocytic, Acute; Leukemia, Myeloid, Acute | interventions — Gemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (monoclonal antibody therapy) (Experimental): Patients receive gemtuzumab ozogamicin IV over 2 hours on days 1 and 15. Treatment continues for 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: gemtuzumab ozogamicin; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: gemtuzumab ozogamicin — Given IV
  Other Names: Calicheamicin-Conjugated Humanized Anti-CD33 Monoclonal Antibody; CDP-771; CMA-676; Mylotarg
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This clinical trial studies the side effects of gemtuzumab ozogamicin and how well it works in treating patients with acute myeloid leukemia. Monoclonal antibodies, such as gemtuzumab ozogamicin, can block cancer growth in different ways. Some block the ability of cancer to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To study safety and efficacy single agent Gemtuzumab Ozogamicin (Mylotarg®) as induction therapy for patients with Acute Myeloid Leukemia (AML) who have relapsed after standard treatments or who are not candidates for standard consolidation treatment after Daunorubicin and cytosine arabinoside.

SECONDARY OBJECTIVES:

I. To correlate morbidity and mortality with the use of gemtuzumab (gemtuzumab ozogamicin) to specific subtypes of leukemia.

II. To correlate gemtuzumab response to degree of cluster of differentiation (CD) 33 positivity.

III. To correlate FMS-Related Tyrosine Kinase 3 (FLT 3)/nucleophosmin (NPM) status and CD 33 positivity to gemtuzumab response.

IV. To document incidence of sinusoidal obstruction syndrome with the use of gemtuzumab.

OUTLINE:

Patients receive gemtuzumab ozogamicin intravenously (IV) over 2 hours on days 1 and 15. Treatment continues for 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up monthly for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have confirmed relapsed or refractory acute myeloid leukemia and not a candidate for standard induction treatment after daunorubicin and cytosine arabinoside OR acute promyelocytic leukemia relapsed after all-trans retinoic acid (ATRA) or Arsenic trioxide therapy
* Patients must have an initial diagnosis of acute myeloid leukemia or biphenotypic acute leukemia
* Patients must have CD33 positivity of >= 30%
* Eastern Cooperative Oncology Group (ECOG) performance status =< 3
* Karnofsky > 60%
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) =< 2 X institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 30 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* The effects of Mylotarg on the developing human fetus are unknown; for this reason and because Mylotarg class agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients may not be receiving any other investigational agents for leukemia
* Patients with known untreated Hepatitis C because veno-occlusive disease and liver enzyme abnormalities have been associated with Mylotarg
* Uncontrolled intercurrent illness including, but not limited to active liver disease, ongoing or active sepsis requiring vasopressors or mechanical ventilation, symptomatic congestive heart failure, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because Mylotarg is a Class D agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with Mylotarg, breastfeeding should be discontinued if the mother is treated with Mylotarg
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with Mylotarg; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* Congestive Heart Failure (CHF) with an ejection fraction < 30%
* Glomerular filtration rate (GFR) < 30ml/min
* Active central nervous system (CNS) involvement of leukemia
* Philadelphia chromosome + acute lymphoblastic leukemia (ALL)
* Prior hematopoietic transplant in last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-05; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Rate of serious adverse events | Approximately 1 year
  95% confidence interval will be calculated. Graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

SECONDARY OUTCOMES:
Overall response, defined as complete remission (CR) and CR with incomplete platelet recovery (CRp) | At 28 days
Safety analysis of gemtuzumab ozogamicin as induction therapy for patients with relapsed AML | Approximately 1 year
  Adverse event frequency and severity
Overall survival (OS) | Approximately 1 year
Event-free survival (EFS) | Approximately 1 year
Disease free survival (DFS) | Approximately 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Ellis, MD, Principal Investigator — Wake Forest University Health Sciences